CLINICAL TRIAL: NCT06413615
Title: A Phase 2, Multicenter, Open-Label Study to Assess the Efficacy, Safety, Tolerability and Pharmacokinetics of FDA022-BB05 in Patients with Advanced/Metastatic Solid Tumors
Brief Title: A Study of FDA022-BB05 in Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F0034-201
Record Dates: First submitted 2024-05-08; First posted 2024-05-14 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-04

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HER2 Low Metastatic/Recurrent Breast Cancer (Experimental): Enrolled Subjects will receive a 5.4 mg/kg IV dose of FDA022-BB05 on Day 1 of each cycle Q3W
  Interventions: Drug: FDA022-BB05
- HER2 Expressing Metastatic/Recurrent Endometrial Cancer (Experimental): Enrolled Subjects will receive a 5.4 mg/kg IV dose of FDA022-BB05 on Day 1 of each cycle Q3W
  Interventions: Drug: FDA022-BB05
- HER2 Overexpressing/Mutant Metastatic/Recurrent Solid tumor (Experimental): Enrolled Subjects will receive a 5.4 mg/kg IV dose of FDA022-BB05 on Day 1 of each cycle Q3W
  Interventions: Drug: FDA022-BB05

INTERVENTIONS:
Drug: FDA022-BB05 — Monoclonal antibody-drug conjugate for injection

SUMMARY:
This is an open-label, multicenter, Phase II study to evaluate the efficacy and safety of FDA022-BB05 for the treatment in locally advanced, unresectable, or metastatic patients with selected HER2 overexpressing/expressing solid tumors which are not eligible for curative therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects fully understand and voluntarily participate in this study and sign informed consent.

Left Ventricular Ejection Fraction (LVEF) ≥ 50% within 28 days prior to first dose.

Eastern Cooperative Oncology Group performance status( PS) of 0 or 1. Life expectancy ≥ 3 months.

Histopathologically or cytologically confirmed advanced/unresectable or metastatic solid malignant tumors that is refractory to or intolerable with standard treatment, or for which no standard treatment is available:

Cohort A: Pathologically documented breast cancer that:

* Is unresectable or metastatic.
* Has a history of low HER2 expression, defined as IHC 2+/ISH- or IHC 1+ (ISH- or untested).
* For HR-positive participants, is documented refractory to endocrine therapy, defined as having progressed on at least 1 endocrine therapy and determined by the investigator that subject would no longer benefit from further treatment from endocrine therapy.
* Was never previously HER2-positive(IHC 3+ or IHC 2+/ISH+) on prior pathology testing or was historically HER2 IHC 0 only.

Cohort B: Pathologically documented endometrial cancer that:

* Is unresectable or metastatic.
* Has a history of HER2 expression, defined as HER2 1+, 2+, or 3+ score on immunohistochemistry (IHC).
* Have had at least one prior line of platinum-based therapy (in any setting).
* Was never previously received other ADC anti-tumor treatment.

Cohort C: Metastatic or advanced solid tumor that are HER2 overexpression or mutation(Including urothelial cancer, colorectal adenocarcinoma and non-small cell lung cancer).

Exclusion Criteria:

* A treatment history of antibody-drug conjugate containing topoisomerase I inhibitors.

Subjects with one of the following conditions prior to first dose, including, but not limiting to：A major operation or severe trauma history within 4 weeks; A history of chemotherapy, targeted therapy, anti-angiogenesis therapy, biotherapy, immunotherapy, radiotherapy or other anti-tumor therapy within 4 weeks; A history of endocrine therapy within 3 weeks; A history of autologous stem cell transplant within 3 months.

Subjects with other malignant tumors in the past three years (not including cured non-melanoma skin basal cell carcinoma, cervical carcinoma in situ and other malignancies of low malignant potential that have been effectively controlled without treatment).

Subjects with symptomatic CNS metastasis (for example, cerebral edema requiring glucocorticoids therapy, or progressive CNS metastasis), not including prior cerebral and meningeal metastasis that is confirmed stable with MRI and without systematic glucocorticoids therapy.

Adverse reactions from the previous anti-tumor treatment have not yet recovered (>Grade 2 in NCI-CTCAE 5.0, with exception of alopecia and pigmentation or other adverse reactions judged no safety risk by the investigator).

Subjects with clinically significant cardiovascular or cerebrovascular disease, including, but not limiting to:

a medical history of symptomatic Congestive Heart Failure (CHF) (NYHA classes II-IV) or serious cardiac arrhythmia.

a medical history of myocardial infarction or unstable angina within 6 months prior to screening; a QTc prolongation to > 450 millisecond (ms) in males and > 470 ms in females.

Subjects with a medical history of interstitial lung disease (ILD)/pneumonia in need of glucocorticoids intervention，or with interstitial lung disease, or suspicious ILD by imaging detection at screening.

Subjects with any uncontrolled active infection within 1 week prior to first dose.

Subjects with concomitant disease potentially increasing toxicological risk. Known allergy to protein preparation or any protein drug with similar structure to FDA022-BB05.

Subjects with a History of alcohol abuse or psychotropic/narcotic drug abuse; Pregnant or lactating women. Subjects with poor compliance, or not suitable for this study as determined by the investigator due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 24 month
  The percentage of patients with CR and PR assessed by investigators according to RECIST v 1.1
Occurrence of adverse events (AEs) and serious adverse events (SAEs) | up to 24 month
  Occurrence of AEs and SAEs graded according to NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Duration of response (DoR) | up to 24 month
  DOR is defined as the time from the date of first documented response until the date of documented progression or death.
Disease control rate (DCR) | up to 24 month
  DCR is the percentage of subjects who have a best overall response of complete response (CR) or partial response (PR) or stable disease (SD).
Progression free survival (PFS) | up to 24 month
  PFS is the time from date of first dose of study treatment until the date of objective disease progression or death.
Overall survival (OS) | up to 24 month
  OS is the time from date of first dose of study treatment until death due to any cause.
Pharmacokinetic (PK) Analysis: Area Under the Concentration Versus Time Curve (AUC) of Serum FDA022-BB05 Following First Dose | From cycle1 to Cycle10 (each cycle is 21 days. )
  The serum PK parameters of FDA022-BB05 and its analytes for area under the concentration-versus-time curve from time 0 to the last quantifiable concentration as calculated by the linear-up log-down trapezoidal method (AUClast) and AUC from time 0 to infinity (AUCinf) elimination rate constant associated with the terminal phase were estimated using standard non-compartmental methods.
Pharmacokinetic Analysis: Maximum (Peak) Observed Serum Concentration (Cmax) of Serum FDA022-BB05 Following First Dose | From cycle1 to Cycle10 (each cycle is 21 days. )
  The serum PK parameters Maximum (peak) Observed serum concentration of FDA022-BB05 and its analytes were estimated using standard non-compartmental method.
Pharmacokinetic Analysis: Time of Maximum Plasma Concentration (Tmax) of Serum FDA022-BB05 Following First Dose | From cycle1 to Cycle10 (each cycle is 21 days. )
  The serum PK parameters of Time of maximum plasma concentration (Tmax) for FDA022-BB05 and its analytes were estimated using standard non-compartmental methods.
Pharmacokinetic Analysis: Terminal Elimination Half-life (t1/2) of Serum FDA022-BB05 Following First Dose | From cycle1 to Cycle10 (each cycle is 21 days. )
  The serum PK parameters of Terminal elimination half-life for FDA022-BB05 and its analytes was estimated using standard non-compartmental methods.
Number of participants who developed measurable anti-drug antibodies | up to 24 month
  Individual participant data and descriptive statistics will be provided for data at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No